CLINICAL TRIAL: NCT05698576
Title: TRANBERG® Transperineal MR/US Focalyx Fusion Laser--Induced Thermal Therapy in the Office Setting Under Local Anesthesia
Brief Title: TRANBERG® Transperineal MR/US Fusion Laser--Induced Thermal Therapy for Men With Prostate Cancer
Acronym: TPF-LITT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Urological Research Network, LLC (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: URN-2022-002; Pro00060491 (Other: ADVARRA IRB)
Record Dates: First submitted 2022-01-19; First posted 2023-01-26 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Prostate Cancer; Adverse Effects Surgery; MRI; Ultrasound; Sexual Function Disturbances; Urinary Incontinence; Urinary Function Disorders; Prostate Biopsy; Ablation
MeSH Terms: conditions — Prostatic Neoplasms; Sexual Dysfunctions, Psychological; Urinary Incontinence

STUDY DESIGN:
Intervention Model Description: Voluntary participation in a Prospective controlled cohort
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- TPF-LITT ARM (Experimental): partial gland ablation of the prostate using laser device and imaging fusion
  Interventions: Device: TRANBERG® Transperineal Fusion Laser--Induced Thermal Therapy of Prostate Cancer (TPF-LITT)

INTERVENTIONS:
Device: TRANBERG® Transperineal Fusion Laser--Induced Thermal Therapy of Prostate Cancer (TPF-LITT) — A perineal local anesthesia block is performed with patient on lithotomy. The ultrasound probe is advanced, secured to digital stepper. The live ultrasound image feed is visible on the FOCALYX® Fusion device. Image co-registration (MR/US) will be performed. The FOCALYX® Fusion device shows outline of the prostate on the MRI and the target area(s) in real-time. The urologist advances laser fiber introducer, temperature probes to indicated coordinates. Target treatment - applying TRANBERG® laser energy over the treatment area and controlling delivery with a pedal. Treatment is monitored using FOCALYX® Fusion device in real-time. One laser fiber will be used and a single or multiple applications may be required. The fiber will be relocated to other targets if present. Patient will be dismissed to the MRI center where a multiparametric MRI will be conducted. After this study is completed, the patient will be discharged home with instructions and contact information.
  Other Names: Fusion Imaging Laser induced thermal therapy for prostate partial gland ablation.

SUMMARY:
This study is set up as a phase I prospective, single center, device interventional pilot study carried in office setting under local anesthesia. It will assess the tolerance and safety of target fusion ablation of prostate cancer tumors using Laser Induced Thermal Therapy (TFA-LITT) guided by fusion imaging in men 50 to 80 years of age with low to intermediate risk prostate cancer

Prostate Cancer is currently managed with in a discrete fashion where patients either enroll in active surveillance protocols (No intervention) or undergo full intervention via whole gland treatments - most commonly radical surgery or radiation. These treatments have not shown definitive gains in all cause survival and not uncommonly harbor undesirable adverse effects, most notably: impotency and incontinence. Such events elicit significant and noticeable changes on a male lifestyle and for most prostate cancer tumors are considered overtreatment. This study aims to evaluate the use of TFA-LITT in the office setting under local anesthesia - greatly decreasing patient perioperative surgical risk - focused on the organ sparing cancer lesion ablation, where organ function is preserved.

The fundamental objective is to determine the tolerance and safety of TFA-LITT in men with low to intermediate risk prostate cancer, successful performed in the outpatient office-based setting under local anesthesia directed by fusion imaging. Secondary objectives include: 1-Biopsy proven cancer control of ablated areas 12 months after procedure; 2-Uroflowmetry and urinary function Patient Reported Outcome Measures (PROMs) at one, three, six, nine and 12 months; 3- Sexual function Patient Reported Outcome Measures (PROMs) at one, three, six, nine and 12 months; 4- MRI changes of ablated area one, three and 12 months after TFA-LITT; 5- Absence or presence of ejaculation after TFA-LITT.

DETAILED DESCRIPTION:
The field of urology currently demands better options for men diagnosed with prostate cancer, the most common solid tumor in the US and Western Europe. Recently, active surveillance has become a main alternative for patients and physicians seeking to avoid the overtreatment phenomenon associated with standard treatments. However, most men on surveillance protocols for prostate cancer end up converting to "definitive" management whether surgery or radiation within 5 years from diagnosis.

The TRANBERG®|Thermal Therapy System (Clinical Laserthermia Systems AB. Scheelevägen 2 | 223 81 Lund, Sweden), is a 25 W, 1064 nm diode laser. It uses a disposable laser applicator 14G that allows the insertion of a laser applicator (15G) with a fiberoptic core of 550µm. This thermal therapy laser system is indicated for minimal invasive ablation procedures so called Laser Induced Thermal Therapy (LITT) or also called Laser Ablation for prostate treatments. During LITT, light causes damage in tissue due to absorption of light and through heat conduction into the tissue of the absorbed energy. Light tissue interaction is reliable, reproducible, and safe. The laser fiber tip induces necrosis near the tip and coagulative effects deeper in tissues through heat conduction. The body cleans up treated tissue over time. Much experience is gained with laser ablation in different organs.

The development of medical fusion devices that incorporate the precise diagnostic findings from MRI with the flexibility of ultrasound has expanded the precision of prostate biopsies and has led thinking into the current management of prostate cancer, opening for consideration the case for partial gland ablation as an option with fewer side effects.12 Conceivably, the most promising role of fusion imaging would be in the management spectrum of prostate cancer. MRI/US fusion imaging has tremendous advantages, it delivers precise anatomical boundaries and perspectives to surgeons as they sought to destroy cancer lesions and spare healthy tissue. A better understanding on their role in ablation treatments is imperative.

The Focalyx® Fusion (Focalyx, 2140 West 68th St, #204a. Miami Lakes, FL, USA) is a novel disruptive medical device that enables an office based transperineal approach to be conducted using real-time fusion. The characteristics of this fusion device and trials studies have been well documented. This theoretically makes available a safe and laser fiber energy delivery that results in expedient and short procedure times. The Focalyx® Fusion has been used safely in the transperineal diagnosis (fusion biopsies) and management (fusion targeted cryoablation) of men with Prostate Cancer in the office setting. However, targeted prostate cryoablation carries some intrinsic disadvantages as it requires high pressure gasses. Argon and helium are not readily available worldwide, and its efficacy depends on several timely cycles demanding procedure times of about an hour or more. LITT can be accomplished in efficient minutes treatment times and can address the multi-focality of prostate cancer quite effectively. Laser ablation has proven effective when conducted in an MRI bore, however, the immensity of these machines, limited size of the bore, prone positioning and constant in and out verification makes this approach not practical. Fusion laser ablation for prostate cancer is a novel concept that can bring together the precision of MRI with the practicality of ultrasound.

The combination of the TRANBERG® laser and the FOCALYX® Fusion medical device will allow us to perform targeted transperineal fusion laser induced thermal therapy (TPF-LITT) of prostate cancer lesions. This approach portends significant advantages that the investigators can consider, among them: lesion directed ablation, sparring of critical organs and structures such as the bladder neck, NVB, urethral sphincter and rectum. Moreover, healthy tissue is spared and can perform its function, if it mirrors what the investigators have accomplished with target fusion cryoablation. It shall be expected that most men will have preservation of some ejaculation, mild changes in sexual function and no incontinence following treatment with TPF-LITT. In fact, from a urinary function status, the investigators expect patients to suffer no harm either subjectively or objectively. However, all these thoughts require rigorous evaluation. Today, there is no data or evaluation of its safety profile if/when conducted in an office setting under local anesthesia. Therefore, in this study, the principal aim is to assess tolerability and safety profile of TRANBERG® TPF-LITT conducted in men with Prostate Cancer in the office setting.

Objective: The primary objective of this study is to assess tolerability and safety, of TRANBERG® TPF-LITT in Prostate Cancer patients with clinically localized disease. The secondary objectives are to evaluate clinical performance, changes in erectile and sexual function as well as imaging volumetric changes in prostate lesions, prostate size as well as cancer control in treated areas Study design: This study is set up as open label, prospective, single center, interventional study.

Study population: Patients with low or intermediate risk prostate cancer ≥ 50 years of age.

Study Intervention: Upon meeting inclusion and exclusion criteria, subjects will undergo prostate ablation planning where the ablation areas will be noted irrespective of location so long, they are confined to this organ. The planning will allow to spare, if possible, critical structures such as the urethra, neurovascular bundles, and bladder neck. TRANBERG® TPF-LITT treatment execution will be conducted under local anesthesia using the FOCALYX® Fusion medical device as guidance for precise laser fiber localization and real-time monitoring. This investigation will employ a single fiber that will be repositioned to destroy several targeted areas to achieve the TFP-LITT goals. The surgeon will deliver the laser energy and adjust if needed. The areas treated will develop coagulative necrosis with scarring as a response to TPF-LITT. Upon conclusion of the procedure, the patient will have a multiparametric MRI of the prostate to determine the extent of ablation with this powerful technology immediately after treatment, and subsequently 1, 3 and 12 months after.

Main study parameters/endpoints: Tolerability and safety represents the main endpoints of this trial. Tolerability will be assessed during the execution of TFP-LITT. Patients will be provided with a pain analog scale and pain scores will be recorded before initiation of the procedure and during several milestones of the procedure. A final overall pain assessment will be recorded as well. Safety will be assessed during the 7-day, 30-day and 90-day clinic visits. Adverse events (AEs) will be monitored and reported using the CTCAE scale, as perioperative assessments will be conducted at each of these milestones. A grade 3 or worse AEs based on the CTCAE v5.0 within 90 days post procedure will be considered severe. Secondary outcomes will include cancer control, urinary and sexual functional outcomes. Cancer control will be measured with MRI at several milestones, serum PSA changes during the year and the definitive measure will be a Transperineal MR/US Fusion Biopsy at one year of follow up. Urinary and Sexual functional outcomes will be determined by evaluating changes in the validated questionnaires. Ejaculation will be monitored by direct questions.

The investigators aim to streamline the follow up focusing on safety according to standard of care. Patients will be instructed to contact us if they perceive any AEs. The principal investigator will oversee each patient for any AEs. Patients will be followed up in the clinic 7 days post procedure for catheter removal and AEs assessments. They will be contacted 30 days after the procedure and an AEs questionnaire will be administered as well. AEs, IPSS and SHIM assessments will be done at the 6 weeks and 3-month visits. IPSS and SHIM assessments will be done at the 6-month, 9-months and 12-months visits. Flow and volumetric studies will be conducted 3 months and 12 months from procedure date. From an oncological perspective, patients will have serum markers evaluations - PSA, Testosterone Creatinine and GFR measurements prior to a multiparametric MRI and subsequently before each MRI at months 1, 3 and 12 after TPF-LITT procedure. Critically, the Focalyx® Fusion device will be used to assess the delta changes for each lesion and overall change in prostate configuration after each MRI performed. This will allow further understanding of the speed of tissue retraction, remodeling, and spatial orientation of the treated areas for each patient. Finally at 12 months, a MR/US Transperineal fusion biopsy will be performed to assess the ablated tissue cancer sterility.

In Conclusion, TRANBERG® TPF-LITT will expose patients to potential intervention risks. However, it is our estimation and bias these potential risks will be favorable or equal to those observed with compared available standard minimal invasive treatment approaches such as active surveillance. The risks usually associated with transrectal procedures is eliminated as all treatments will performed via a transperineal access. The burden is in our opinion favorable and acceptable.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to sign informed consent
* Subject is able and willing to complete all procedure and follow-up visits indicated in the protocol
* Absence of urinary retention
* Prostate volume: ≥ 18 and ≤ 100 cc, measured by transrectal ultrasound
* Serum creatinine levels <2 ng/dl and GFR > 45
* Serum PSA levels < 20 ng/ml
* Multiparametric prostate MRI with piRADS scores 3-5
* Prostate volume: ≥ 18 and ≤ 100 cc, measured by MRI
* Presence of Intermediate risk prostate cancer with a volume that is less than 1/3 of the gland volume by MRI evaluation

Exclusion Criteria:

* Post-void residual (PVR): > 250 mL or > 50% of voided volume
* Previous prostate cancer intervention (Radiation therapy, brachytherapy, prostate cryoablation
* Major neurological conditions such as Alzheimer's, Parkinson, Multiple sclerosis, ALS, spinal cord injury
* Evidence of neurogenic bladder determined by urodynamics studies
* Presence of Indwelling Foley catheter or on active regime of clean intermittent catheterization (CIC) in the prior 30 days
* Active urinary tract infection determined by urinary cultures
* SHIM score <14
* IPSS score >23
* Acute prostatitis
* Macroscopic hematuria without a known contributing factor
* History of colorectal carcinoma with anterior perineal resection of rectum
* History of pelvic radiation therapy or radical pelvic surgery
* History of bladder neck contracture and/or urethral strictures within the 5 years prior to the informed consent date
* Bladder stones
* Medical contraindication for undergoing TPFLA surgery (eg, infection, coagulopathy, significant cardiac or other medical risk factors for surgery)
* Diagnosed or suspected bleeding or coagulopathic disorder such as hemophilia, ITP, TTP
* Medical contraindication to being subjected to local anesthesia

Ages: 50 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-03-16 (Actual); Primary Completion 2023-01-27 (Estimated); Study Completion 2033-01-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] of TRANBERG® TPF-LITT performed in the office setting under local anesthesia. | 90 days
  Tolerability will be assessed during the execution of TFP-LITT at several phases of the treatment. An analog pain scale will be provided to the patient, whom will be asked to describe any pain scores at each of the following treatment successions:
  1. superficial perineal block,
  2. foley advancement,
  3. deep perineal block,
  4. fusion co-registration,
  5. before and after each ablation, 6-Once the patient has recovered, he will be asked for an overall pain assessment.
  Safety will be evaluated by assessments of the 7-day, 30-day and 90-day AEs reported using the CTCAE scale, as perioperative assessments will be conducted at each of these milestones. A grade 3 or worse AEs based on the CTCAE v5.0 within 90 days post procedure will be considered severe. Any registered AEs will be labelled as follows:
  1. Not related
  2. Possible
  3. Probable
  4. Causal relationship

SECONDARY OUTCOMES:
Average Ablated area volume (in cc) measured by MRI immediately following the procedure | 24-72 hours after procedure
  patients will undergo a multiparametric MRI immediately after the procedure and the ablated areas will be contoured and the dimensions on cubic centimeters will be recorded as ablation area
Average Ablated area volume (in cc) measured by MRI 1-month following the procedure | 30 days
  patients will undergo a multiparametric MRI 30 days (1-month) after the procedure and the ablated areas will be contoured and the dimensions on cubic centimeters will be recorded as ablation area
Average Ablated area volume (in cc) measured by MRI 3-month following the procedure | 90 days
  patients will undergo a multiparametric MRI 90 days (3-month) after the procedure and the ablated areas will be contoured and the dimensions on cubic centimeters will be recorded as ablation area
Average Ablated area volume (in cc) measured by MRI 1-year following the procedure | 1 year
  patients will undergo a multiparametric MRI 1-year after the procedure and the ablated areas will be contoured and the dimensions on cubic centimeters will be recorded as ablation area
Number of patients with a 75% decrease in Serum PSA levels (ng/ml) after procedure measured at fixed intervals | 1 year
  The PSA will be obtained as well at 1, 3, 6, 9 and 12-months post procedure.
Number of patients with presence of cancer cells in treated -ablated- area | 1 year
  pathological assessment of samples obtained trough a MR/US Transperineal Fusion biopsy of the prostate treated area
Number of patients with a 50% increase in qMAX measured in cc/second on flow studies | 12 Months
  Uroflowmetry in cc/s will be performed on patients at 3 and 12 months after the procedure. Assessment of maximal flow rate -qmax (cc/seconds) will be obtained
Number of patients with a 7 point drop in the International Prostate Symptom Score (IPSS) | 12 Months
  Patients will be asked to answer the validated questionnaire - international prostate symptom scores (IPSS) - at 1,3 ,6 ,9 and 12 months following the procedure The IPSS scores range from 1 to 35
Number of patients with a 5 point drop in the sexual health inventory for men (SHIM) scores | 12 Months
  Patients will be asked to answer the validated questionnaire - sexual health inventory for men (SHIM) - at 1,3 ,6 ,9 and 12 months following the procedure The SHIM scores range from 1 to 25
Number of men with absent ejaculation | 12 Months
  Assessed by a direct yes or no answer to the question at 1,3 ,6 ,9 and 12 months following the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Fernando J Bianco, MD, Principal Investigator — Urological Research Network; Isabel H Lopez, BS., MBA, Study Director — Urological Research Network
Locations (1):
- Urology Specialist Group, Hialeah, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
De-Identified datasets may be shared for Meta-Analysis purposes or Matched cohort analysis
Supporting Information: CSR
Time Frame: 3 years
Access Criteria: formal request, institutional agreements

REFERENCES:
- [Background] Carter G, Clover K, Britton B, Mitchell AJ, White M, McLeod N, Denham J, Lambert SD. Wellbeing during Active Surveillance for localised prostate cancer: a systematic review of psychological morbidity and quality of life. Cancer Treat Rev. 2015 Jan;41(1):46-60. doi: 10.1016/j.ctrv.2014.11.001. Epub 2014 Nov 13. PMID 25467109
- [Background] Cooperberg MR, Carroll PR, Klotz L. Active surveillance for prostate cancer: progress and promise. J Clin Oncol. 2011 Sep 20;29(27):3669-76. doi: 10.1200/JCO.2011.34.9738. Epub 2011 Aug 8. PMID 21825257
- [Background] Hamdy FC, Donovan JL, Lane JA, Mason M, Metcalfe C, Holding P, Davis M, Peters TJ, Turner EL, Martin RM, Oxley J, Robinson M, Staffurth J, Walsh E, Bollina P, Catto J, Doble A, Doherty A, Gillatt D, Kockelbergh R, Kynaston H, Paul A, Powell P, Prescott S, Rosario DJ, Rowe E, Neal DE; ProtecT Study Group. 10-Year Outcomes after Monitoring, Surgery, or Radiotherapy for Localized Prostate Cancer. N Engl J Med. 2016 Oct 13;375(15):1415-1424. doi: 10.1056/NEJMoa1606220. Epub 2016 Sep 14. PMID 27626136
- [Background] Loeb S, Carter HB, Schwartz M, Fagerlin A, Braithwaite RS, Lepor H. Heterogeneity in active surveillance protocols worldwide. Rev Urol. 2014;16(4):202-3. No abstract available. PMID 25548550
- [Background] Cooley LF, Emeka AA, Meyers TJ, Cooper PR, Lin DW, Finelli A, Eastham JA, Logothetis CJ, Marks LS, Vesprini D, Goldenberg SL, Higano CS, Pavlovich CP, Chan JM, Morgan TM, Klein EA, Barocas DA, Loeb S, Helfand BT, Scholtens DM, Witte JS, Catalona WJ; Collaborators. Factors Associated with Time to Conversion from Active Surveillance to Treatment for Prostate Cancer in a Multi-Institutional Cohort. J Urol. 2021 Nov;206(5):1147-1156. doi: 10.1097/JU.0000000000001937. Epub 2021 Sep 10. PMID 34503355
- [Background] Al-Hakeem Y, Raz O, Gacs Z, Maclean F, Varol C. Magnetic resonance image-guided focal laser ablation in clinically localized prostate cancer: safety and efficacy. ANZ J Surg. 2019 Dec;89(12):1610-1614. doi: 10.1111/ans.15526. Epub 2019 Nov 3. PMID 31679182
- [Background] Lee T, Mendhiratta N, Sperling D, Lepor H. Focal laser ablation for localized prostate cancer: principles, clinical trials, and our initial experience. Rev Urol. 2014;16(2):55-66. PMID 25009445
- [Background] Walser E, Nance A, Ynalvez L, Yong S, Aoughsten JS, Eyzaguirre EJ, Williams SB. Focal Laser Ablation of Prostate Cancer: Results in 120 Patients with Low- to Intermediate-Risk Disease. J Vasc Interv Radiol. 2019 Mar;30(3):401-409.e2. doi: 10.1016/j.jvir.2018.09.016. PMID 30819483
- [Background] Kasivisvanathan V, Rannikko AS, Borghi M, Panebianco V, Mynderse LA, Vaarala MH, Briganti A, Budaus L, Hellawell G, Hindley RG, Roobol MJ, Eggener S, Ghei M, Villers A, Bladou F, Villeirs GM, Virdi J, Boxler S, Robert G, Singh PB, Venderink W, Hadaschik BA, Ruffion A, Hu JC, Margolis D, Crouzet S, Klotz L, Taneja SS, Pinto P, Gill I, Allen C, Giganti F, Freeman A, Morris S, Punwani S, Williams NR, Brew-Graves C, Deeks J, Takwoingi Y, Emberton M, Moore CM; PRECISION Study Group Collaborators. MRI-Targeted or Standard Biopsy for Prostate-Cancer Diagnosis. N Engl J Med. 2018 May 10;378(19):1767-1777. doi: 10.1056/NEJMoa1801993. Epub 2018 Mar 18. PMID 29552975
- [Background] Simmons LAM, Kanthabalan A, Arya M, Briggs T, Barratt D, Charman SC, Freeman A, Gelister J, Hawkes D, Hu Y, Jameson C, McCartan N, Moore CM, Punwani S, Ramachandran N, van der Meulen J, Emberton M, Ahmed HU. The PICTURE study: diagnostic accuracy of multiparametric MRI in men requiring a repeat prostate biopsy. Br J Cancer. 2017 Apr 25;116(9):1159-1165. doi: 10.1038/bjc.2017.57. Epub 2017 Mar 28. PMID 28350785
- [Background] Bianco FJ, Martinez-Salamanca JI. Focalyx Dx, Bx, Tx et Apps: A novel contemporary fusion paradigm for the management of prostate cancer. Arch Esp Urol. 2016 Jul;69(6):353-63. PMID 27416639
- [Background] Hu Y, van den Boom R, Carter T, Taylor Z, Hawkes D, Ahmed HU, Emberton M, Allen C, Barratt D. A comparison of the accuracy of statistical models of prostate motion trained using data from biomechanical simulations. Prog Biophys Mol Biol. 2010 Dec;103(2-3):262-72. doi: 10.1016/j.pbiomolbio.2010.09.009. Epub 2010 Sep 30. PMID 20869389
- See also: PROPHYLACTIC ANTIBIOTICS IN TRANSPERINEAL PROSTATE BIOPSIES. ARE THEY REALLY NECESSARY? Fernando Bianco, Eusebio Luna, Alberto Lopez-Prieto, Farshad Shafizadeh, Hu Jim, Edward Gheiler, Ariel Kaufman, Juan Martinez-Salamanca, Luanda Y. Perez, Barrios D — http://doi.org/10.1097/JU.0000000000002023.03